CLINICAL TRIAL: NCT04355962
Title: Sevoflurane Sedation in COVID-19 ARDS Patients to Reduce Lung Injury: a Randomized Controlled Trial
Brief Title: Sevoflurane in COVID-19 ARDS (SevCov)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Kantonsspital Münsterlingen (Other); Triemli Hospital (Other); Cantonal Hospital of St. Gallen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-00719
Record Dates: First submitted 2020-03-26; First posted 2020-04-21 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: ARDS, Human; Coronavirus
Keywords: COVID-19; ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome; Coronavirus Infections; COVID-19 | interventions — Sevoflurane; Infusion Pumps

STUDY DESIGN:
Intervention Model Description: a randomized, controlled multi-center trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not be informed about their group assignments, technicians processing the samples will not have any access to the ICU or the patient chart (= double-blind trial). Due to the procedures involved in volatile versus intravenous sedation, group assignment cannot be entirely concealed for the study staff and ICU doctors/nurses involved with the procedure in the ICU (pragmatic limits of blinding).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane Sedation (Experimental): Sedation with sevoflurane (etSevo 0.5-1.5 Vol %) for 48 hours in patients with COVID-19 ARDS
  Interventions: Drug: Sevoflurane
- Intravenous (Active Comparator): No use of sevoflurane, but current intravenous sedation at discretion of the ICU physician in charge, e.g. with propofol, fentanyl, midazolam and dexmedetomidine
  Interventions: Drug: Intravenous drug

INTERVENTIONS:
Drug: Sevoflurane — Sedation with sevoflurane (etSevo 0.5-1.5 Vol %) for 48 hours in patients with COVID-19 ARDS
  Arms: Sevoflurane Sedation
Drug: Intravenous drug — Intravenous sedation in control group will be continued as initiated at the ICU e.g. propofol, fentanyl, midazolam, dexmedetomidine
  Arms: Intravenous

SUMMARY:
The purpose of this trial is to study the effect of initial temporary sevoflurane sedation on mortality and persistent organ dysfunction (POD) in survivors at day 28 after ICU admission in the population of patients suffering from COVID-19 ARDS.

DETAILED DESCRIPTION:
The corona virus disease 19 (COVID-19) pandemic, caused by the severe acute respiratory syndrome corona virus 2 (SARS-CoV-2), is spreading rapidly across Europe. While data from European centers are still missing, several publications from Chinese centers are available. Respiratory failure from acute respiratory distress syndrome (ARDS) is the leading cause of mortality, and may be caused or exacerbated by a 'cytokine storm syndrome'.

Recent trials from our group demonstrated that the volatile anesthetic sevoflurane administered during ventilation of patients has anti-inflammatory properties. Moreover, in in vivo studies volatile anesthetics reduce the severity of ARDS compared to intravenous sedation, which has been confirmed in a clinical pilot trial. Attenuating ARDS and thereby improving oxygenation strongly decreases morbidity and mortality of patients.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection (positive testing) or computed tomography (CT) scan-suspected COVID-19 ARDS
* Male and female patients, age 18 to 85 years
* ICU patients with ARDS defined as PaO2/FiO2 < 200mmHg (=26.6kPa)
* Time of intubation not longer than 24 hours
* QTc Time (ECG) not longer than 470 ms ♂ (male)/ 480 ms ♀ (female)
* Sedation and mechanical ventilation in ICU
* Informed consent, signed by a representative or by an independent physician

Exclusion Criteria:

* High dose systemic corticosteroids in the phase before hospitalization (> 10mg/d prednisone or equivalent dose)
* Significant concomitant disease (acute cerebral vascular event, acute coronary syndrome, seizure, burn, neuromuscular disease)
* Organ transplant
* AIDS
* Pregnancy and/or breastfeeding
* Use of cytokine absorber

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Composite outcome of death rate (rate of patients that did not survive) and organ failure rate (rate of patients surviving with persistent organ dysfunction) at day 28 | 28 days
  The effect of sevoflurane application on mortality (rate of patients that does not survive 28 days) and persistent organ dysfunction (rate of patients surviving with a persistent organ failure at day 28) will be assessed. Organ failures are defined as pulmonary failure (necessity of ventilation); cardiovascular failure (need of vasopressors), retail failure (need of renal replacement therapy)

SECONDARY OUTCOMES:
Length of stay ICU | 28 days
  The effect of sevoflurane application on the length of stay at ICU will be determined.
Plasma Inflammatory markers | 8 days
  The impact of sevoflurane on the course of inflammatory markers will be evaluated (pro-calcitonin, PCT; c-reactive protein, CRP; interleukin 6, IL-6; monocyte chemoattractant protein 1, MCP-1)
Length of stay at hospital | 28 days
  The effect of sevoflurane application on the length of stay at hospital will be determined.
Sex-related differences in complications | 28 days
  Sex-related differences in complications will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Beck Schimmer, Prof, Study Chair — University of Zurich
Locations (4):
- Switzerland (4):
  - Kantonsspital Münsterlingen, Münsterlingen
  - Cantonal Hospital of St. Gallen, Sankt Gallen
  - Stadtspital Triemli, Zurich
  - University Hospital Zuirch, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Xie J, Tong Z, Guan X, Du B, Qiu H, Slutsky AS. Critical care crisis and some recommendations during the COVID-19 epidemic in China. Intensive Care Med. 2020 May;46(5):837-840. doi: 10.1007/s00134-020-05979-7. Epub 2020 Mar 2. No abstract available. PMID 32123994
- [Background] Suter D, Spahn DR, Blumenthal S, Reyes L, Booy C, Z'graggen BR, Beck-Schimmer B. The immunomodulatory effect of sevoflurane in endotoxin-injured alveolar epithelial cells. Anesth Analg. 2007 Mar;104(3):638-45. doi: 10.1213/01.ane.0000255046.06058.58. PMID 17312223
- [Background] Yue T, Roth Z'graggen B, Blumenthal S, Neff SB, Reyes L, Booy C, Steurer M, Spahn DR, Neff TA, Schmid ER, Beck-Schimmer B. Postconditioning with a volatile anaesthetic in alveolar epithelial cells in vitro. Eur Respir J. 2008 Jan;31(1):118-25. doi: 10.1183/09031936.00046307. Epub 2007 Sep 26. PMID 17898018
- [Derived] Beck-Schimmer B, Schadde E, Pietsch U, Filipovic M, Dubendorfer-Dalbert S, Fodor P, Hubner T, Schuepbach R, Steiger P, David S, Kruger BD, Neff TA, Schlapfer M. Early sevoflurane sedation in severe COVID-19-related lung injury patients. A pilot randomized controlled trial. Ann Intensive Care. 2024 Mar 27;14(1):41. doi: 10.1186/s13613-024-01276-4. PMID 38536545